CLINICAL TRIAL: NCT03208400
Title: Exposure Treatment in Anxiety Disorders: Proof of Principle for an a Priori Response Prediction Approach
Brief Title: Virtual Reality Exposure in Spider Phobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Julius-Maximilians University (Other)
Collaborators: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Ulrike Lueken, Prof. Dr., Julius-Maximilians University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Spider_VR
Record Dates: First submitted 2017-06-28; First posted 2017-07-05 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Specific Phobia; Cognitive-behavioral Therapy; Virtual Reality
MeSH Terms: conditions — Phobia, Specific | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- virtual reality exposure (Other): one-session exposure conveyed via virtual reality technology
  Interventions: Behavioral: virtual reality exposure

INTERVENTIONS:
Behavioral: virtual reality exposure — one-session exposure conveyed via virtual reality technology

SUMMARY:
While knowledge on the neurobiological signatures of fear and anxiety disorders and, in particular, their association with treatment outcome is accumulating, clinical translation still awaits empirical proof of evidence. Exposure-based cognitive-behavioral therapy (CBT) is a first-line treatment, but clinically significant change is only seen in approx. 50-65% of patients. Patient stratification is a powerful option to increase treatment response; however, developing prognostic markers suitable for single-patient predictions still is in its infancy and crucially requires external cross-validation embedded within an a priori prediction approach - a procedure yet largely missing in the field of biomarker research. Employing a bicentric strategy the aim of this study is to test the hypothesis that a priori prediction of treatment outcome based on neurobiological measures is possible in a second, independent sample. Building upon findings from previous mechanistic studies, These will be incorporated into the development of a predictive pattern comprising fear-relevant genotypes and molecules targeting neuropeptides, related epigenetic signatures as well as neurofunctional activation patterns associated with fear circuitry functions, and clinical data. Pre-treatment neurobiological signatures will be tested for their potential as a predictive response marker towards behavioral exposure (virtual reality exposure treatment (VRET) and an in vivo behavioral avoidance test) in a model disorder of fear circuitry dysfunctions (spider phobia). Multivariate pattern analyses employing a machine learning framework will be used to generate predictions on the individual patient level and to cross-validate markers in a second, independent sample. While at site A predictions will be generated following completion of the treatment, response will be predicted at site B a priori, but in a double-blind manner. Comparison of observed vs. predicted response rates will serve as a test of hypothesis. In addition, neuroplastic (on a subsample) and epigenetic changes induced by VRET treatment will be assessed following treatment and, in case of epigenetics, also after 6-months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* specific phobia (animal subtype: spider phobia) according to criteria of the Diagnostic and Statistical Manual of Mental Disorders, 5th Version (DSM-5)
* right-handedness
* Caucasian descent
* willingness to participate in massed exposure

Exclusion Criteria:

* patients exhibiting a primary other anxiety disorder (panic disorder, agoraphobia, social phobia, generalized anxiety disorder), acute suicidality, psychotic, bipolar I, obsessive-compulsive disorder, posttraumatic stress disorder, severe major depression, borderline personality disorder or substance dependency (except nicotine)
* patients fulfilling MRI-related exclusion criteria
* patients with current pharmacological or psychotherapeutic treatment, as well as those already previously treated with exposure-based CBT
* pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Spider Phobia Questionnaire (SPQ) | 4 weeks
  Change in spider phobia symptoms before (baseline) to after therapy

SECONDARY OUTCOMES:
Behavioral Avoidance Text (BAT) | 4 weeks
  Change (in cm) in the extend to which a living spider can be approached from before to after therapy
Behavioral Avoidance Text (BAT) | 6 months
  Change (in cm) in the extend to which a living spider can be approached from before vs. after 6 month follow-up period
Clinical Global Impressions (CGI) | 4 weeks
  Clinician rated symptom severity after completion of treatment (4 weeks)
Clinical Global Impressions (CGI) | 6 month
  Clinician rated symptom severity after 6 month follow-up period
Spider Phobia Questionnaire (SPQ) | 6 months
  Change in spider phobia symptoms before (baseline) vs. after 6 month follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Lueken, Prof. Dr., Principal Investigator — University Hospital of Wuerzburg
Locations (2):
- Germany (2):
  - Center of Mental Health, Dept. of Psychiatry, Psychosomatics, and Psychiatry, University Hospital of Wuerzburg, Würzburg, Bavaria
  - Dept. of Psychiatry, University Hospital Münster, Münster, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwarzmeier H, Leehr EJ, Bohnlein J, Seeger FR, Roesmann K, Gathmann B, Herrmann MJ, Siminski N, Junghofer M, Straube T, Grotegerd D, Dannlowski U. Theranostic markers for personalized therapy of spider phobia: Methods of a bicentric external cross-validation machine learning approach. Int J Methods Psychiatr Res. 2020 Jun;29(2):e1812. doi: 10.1002/mpr.1812. Epub 2019 Dec 8. PMID 31814209
- [Derived] Chavanne AV, Meinke C, Langhammer T, Roesmann K, Boehnlein J, Gathmann B, Herrmann MJ, Junghoefer M, Klahn L, Schwarzmeier H, Seeger FR, Siminski N, Straube T, Dannlowski U, Lueken U, Leehr EJ, Hilbert K. Individual-Level Prediction of Exposure Therapy Outcome Using Structural and Functional MRI Data in Spider Phobia: A Machine-Learning Study. Depress Anxiety. 2023 Aug 22;2023:8594273. doi: 10.1155/2023/8594273. eCollection 2023. PMID 40224607
- [Derived] Langhammer T, Hilbert K, Adolph D, Arolt V, Bischoff S, Bohnlein J, Cwik JC, Dannlowski U, Deckert J, Domschke K, Evens R, Fydrich T, Gathmann B, Hamm AO, Heinig I, Herrmann MJ, Hollandt M, Junghoefer M, Kircher T, Koelkebeck K, Leehr EJ, Lotze M, Margraf J, Mumm JLM, Pittig A, Plag J, Richter J, Roesmann K, Ridderbusch IC, Schneider S, Schwarzmeier H, Seeger F, Siminski N, Straube T, Strohle A, Szeska C, Wittchen HU, Wroblewski A, Yang Y, Straube B, Lueken U. Resting-state functional connectivity in anxiety disorders: a multicenter fMRI study. Mol Psychiatry. 2025 Apr;30(4):1548-1557. doi: 10.1038/s41380-024-02768-2. Epub 2024 Oct 4. PMID 39367057
- [Derived] Roesmann K, Leehr EJ, Bohnlein J, Gathmann B, Herrmann MJ, Junghofer M, Schwarzmeier H, Seeger FR, Siminski N, Straube T, Dannlowski U, Lueken U. Mechanisms of action underlying virtual reality exposure treatment in spider phobia: Pivotal role of within-session fear reduction. J Anxiety Disord. 2023 Dec;100:102790. doi: 10.1016/j.janxdis.2023.102790. Epub 2023 Oct 14. PMID 37879242